CLINICAL TRIAL: NCT05318001
Title: Investigation of Normative Values of Trimester-Specific Biomechanical and Viscoelastic Properties of Plantar Fascia in Pregnant Women-Pilot Study
Brief Title: Biomechanical and Viscoelastic Properties of Plantar Fascia in Pregnant Women-Pilot Study
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 21
Record Dates: First submitted 2022-03-12; First posted 2022-04-08 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Pregnant Women
Keywords: stiffness; creep; normative data; plantar fascia; pregnant women

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First trimester pregnant women (first pregnancy): This group will consist of women in the first trimester and in first trimester of pregnancy
  Interventions: Other: Evaluation of biomechanics and viscoelastic properties of plantar fascia; Other: Evaluation of Foot Morphological Characteristics; Other: Evaluation of navıcular mobility; Other: Evaluation of Foot Posture
- Second trimester pregnant women (first pregnancy): This group will consist of women in the second trimester and in first trimester of pregnancy
  Interventions: Other: Evaluation of biomechanics and viscoelastic properties of plantar fascia; Other: Evaluation of Foot Morphological Characteristics; Other: Evaluation of navıcular mobility; Other: Evaluation of Foot Posture
- Third trimester pregnant women (first pregnancy): This group will consist of women in the third trimester and in first trimester of pregnancy
  Interventions: Other: Evaluation of biomechanics and viscoelastic properties of plantar fascia; Other: Evaluation of Foot Morphological Characteristics; Other: Evaluation of navıcular mobility; Other: Evaluation of Foot Posture

INTERVENTIONS:
Other: Evaluation of biomechanics and viscoelastic properties of plantar fascia — The biomechanical (Tone-Hz, Stiffness-N/m and decrement) and viscoelastic (creep and relaxation time-ms) properties of the plantar fascia will be measured in the side lying position.
  Measurements will be made with the ankle in neutral position.
Other: Evaluation of Foot Morphological Characteristics — Foot length and width will be measured.
Other: Evaluation of navıcular mobility — The amount of navicular drop of both feet will be measured.
Other: Evaluation of Foot Posture — Foot posture will be evaluated according to Foot Posture Index.

SUMMARY:
The feet, which are support surfaces, are adapted to the physiological relaxation and biomechanical changes that occur during pregnancy. In this adaptation, it has not been objectively clarified how the plantar fascia, which plays a very important role in maintaining the height of the plantar arch, undergoes a change. Therefore, the aim of this pilot study is to investigate the normative values of trimester-specific biomechanical and viscoelastic properties of the plantar fascia, which adapts to changes in foot structure during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* First-time pregnancy
* They are between the ages of 18-40
* Pre-pregnancy Body-Mass-Index (BMI) < 30 kg/m2

Exclusion Criteria:

* Presence of any connective tissue disease that would affect the biomechanical or viscoelastic properties of the fascia
* Deterioration of skin integrity in measurement areas
* Presence of orthopedic, neurological, rheumatic problems that may cause musculoskeletal disorders and deviations from normal in biomechanical alignment
* History of surgery or fracture in the lower extremity and foot-ankle region in the last 6 months
* Defining metabolic disorders such as type I, II diabetes, gestational diabetes mellitus (GDM), preeclampsia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women in the first pregnancy
Study Population: Pregnant women in the first- trimester, second trimester or third trimester (first-time pregnancy)
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of biomechanical properties of plantar fascia | The measurement of the baseline stiffness values of plantar fascia between 10-14 weeks, between 20-24 weeks and between 32-36 weeks.
  Measuring of the stiffness (N/m) of the plantar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the side lying position.
Evaluation of biomechanical properties of plantar fascia | The measurement of the baseline decrement values of plantar fascia between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Measuring of the decrement of the plantar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the side lying position.
Evaluation of biomechanical properties of plantar fascia | The measurement of the baseline tone values of plantar fascia between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Measuring of the tone (Hz) of the plantar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the side lying position.
Evaluation of viscoelastic properties of plantar fascia | The measurement of the baseline creep values of plantar fascia between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Measuring of the creep of the plantar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the side lying position.
Evaluation of viscoelastic properties of plantar fascia | The measurement of the baseline relaxation time values of plantar fascia between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Measuring of the relaxation time (ms) of the plantar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the side lying position.

SECONDARY OUTCOMES:
Evaluation of Body Weight | The measurement of the baseline body weight between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Body weight (kg) will be measured
Evaluation of Body Mass Index (BMI) | The measurement of the baseline BMI between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  BMI will be calculated as person's weight in kilograms divided by the square of height in meters
Evaluation of Foot Morphological Characteristics | The measurement of the baseline foot width between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Foot width (cm) will be measured
Evaluation of Foot Morphological Characteristics | The measurement of the baseline foot length between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Foot length (cm) will be measured
Evaluation of foot mobility | The measurement of the baseline navicular drop values between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Navicular drop values will be measured
Evaluation of foot posture | The measurement of the baseline foot posture characteristics between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Foot posture will be evaluated according to foot posture index.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Challis JR, Lockwood CJ, Myatt L, Norman JE, Strauss JF 3rd, Petraglia F. Inflammation and pregnancy. Reprod Sci. 2009 Feb;16(2):206-15. doi: 10.1177/1933719108329095. PMID 19208789
- [Result] Cherni Y, Desseauve D, Decatoire A, Veit-Rubinc N, Begon M, Pierre F, Fradet L. Evaluation of ligament laxity during pregnancy. J Gynecol Obstet Hum Reprod. 2019 May;48(5):351-357. doi: 10.1016/j.jogoh.2019.02.009. Epub 2019 Feb 20. PMID 30794956
- [Result] Segal NA, Boyer ER, Teran-Yengle P, Glass NA, Hillstrom HJ, Yack HJ. Pregnancy leads to lasting changes in foot structure. Am J Phys Med Rehabil. 2013 Mar;92(3):232-40. doi: 10.1097/PHM.0b013e31827443a9. PMID 23117270
- [Result] Huang J, Qin K, Tang C, Zhu Y, Klein CS, Zhang Z, Liu C. Assessment of Passive Stiffness of Medial and Lateral Heads of Gastrocnemius Muscle, Achilles Tendon, and Plantar Fascia at Different Ankle and Knee Positions Using the MyotonPRO. Med Sci Monit. 2018 Oct 23;24:7570-7576. doi: 10.12659/MSM.909550. PMID 30352050
- [Result] Sanjana F, Chaudhry H, Findley T. Effect of MELT method on thoracolumbar connective tissue: The full study. J Bodyw Mov Ther. 2017 Jan;21(1):179-185. doi: 10.1016/j.jbmt.2016.05.010. Epub 2016 Jun 3. PMID 28167175